CLINICAL TRIAL: NCT04474210
Title: An Open-Label, Single-Dose Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of JNJ-56136379 in Adult Participants
Brief Title: A Study to Evaluate the Effect of Renal Impairment on JNJ-56136379 in Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108802; 56136379HPB1010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Renal Insufficiency
Keywords: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — JNJ-56136379

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Group 1 (Experimental): Participants with severe renal impairment and/or kidney failure (estimated glomerular filtration rate [eGFR] less than [<] 30 milliliter[mL]/minute but not yet on hemodialysis) will receive a single oral dose of JNJ-56136379.
  Interventions: Drug: JNJ-56136379
- Part A: Group 2 (Active Comparator): Healthy participants with normal renal function (eGFR greater than or equal to [>=] 90 mL/minute), will receive a single oral dose of JNJ-56136379.
  Interventions: Drug: JNJ-56136379
- Part B: Group 3 (Optional) (Experimental): Participants with mild renal impairment (eGFR: 60 to 89 mL/minute) will receive a single oral dose of JNJ-56136379.
  Interventions: Drug: JNJ-56136379
- Part B: Group 4 (Optional) (Experimental): Participants with moderate renal impairment (eGFR: 30 to 59 mL/minute) will receive a single oral dose of JNJ-56136379.
  Interventions: Drug: JNJ-56136379
- Part B: Group 5 (Optional) (Experimental): Participants with kidney failure (eGFR: <15 mL/minute and on hemodialysis; pharmacokinetic [PK] to be evaluated during non-dialysis days) will receive a single oral dose of JNJ-56136379.
  Interventions: Drug: JNJ-56136379

INTERVENTIONS:
Drug: JNJ-56136379 — Participants will receive JNJ-56136379 tablets orally.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of a single oral dose of JNJ-56136379 in adult participants with renal impairment compared with healthy participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

- Body mass index (BMI) (kilograms [kg]/height [m]^2) between 18.0 and 38.0 kilogram/meter^2 (kg/m2) (inclusive), and body weight not less than (<) 50 kg

Participants with normal renal function:

* Have normal renal function defined as estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 90 milliliter/minute computed with the online calculator on the CKD-EPI website by use of the Chronic Kidney Disease Epidemiology Collaboration creatinine clearance (CKD-EPIcr) result
* Must have stable renal function as defined as: (a) for participants with impaired renal function: <20 percent (%) change in serum creatinine concentrations between screening and Day -1; (b) for healthy participants: a change in serum creatinine concentration <0.2 milligram per deciliter (mg/dL) between screening and Day -1

Participants with renal impairment:

* Have an impaired renal function based on eGFR as(eGFR computed with the online calculator on the CKD-EPI website providing eGFR (in mL/min units) by use of the CKD-EPIcr result: (a) eGFR <90 to 60 mL/minute for participants in Group 3 (mild renal impairment cohort); (b) eGFR 30 to 59 mL/minute for participants in Group 4 (moderate renal impairment cohort); (c) eGFR <30 mL/minute but not yet on hemodialysis, for participants in Group 1 (severe renal impairment and/or kidney failure); (d) eGFR <15 mL/minute and on hemodialysis, for participants in Group 5 (kidney failure)
* Concomitant medications to treat underlying disease states or medical conditions related to renal impairment are allowed. Participants must be on a stable dose of medication and/or treatment regimen for at least 2 months (3 months for thyroid hormone replacement therapy [HRT]) before dosing as well as during the study

Exclusion Criteria:

- Individuals who take creatine supplements, have a non-standard muscle mass such as amputation, malnutrition, or muscle wasting; because these factors are not accounted for in the prediction equations for GFR chronic kidney disease epidemiology collaboration (CKD EPI)

Participants with normal renal function:

* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or Day -1, as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, body temperature, or 12 lead ECG at screening or Day -1, as deemed appropriate by the investigator

Participants with renal impairment:

* Evidence of clinically apparent concurrent disease based upon complete clinical laboratory testing, full physical examination, or medical history, except for controlled hypertension and those problems directly associated with the primary diagnosis of renal impairment
* Any clinically significant laboratory abnormality except abnormalities that may be caused by renal impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) | Up to Day 29
  Cmax is defined as the maximum observed plasma analyte concentration.
Time to Reach the Maximum Observed Plasma Analyte Concentration (Tmax) | Up to Day 29
  Tmax is defined as the actual sampling time to reach the maximum observed plasma analyte concentration.
Area Under the Analyte Concentration-time Curve From Time Zero to 24 Hours Postdose (AUC [0-24]) | Up to 24 hours postdose
  AUC (0-24) is defined as area under the analyte concentration-time curve (AUC) from time 0 to 24 hours postdose, calculated by linear-linear trapezoidal summation.
Area Under the Analyte Concentration-time Curve From Time Zero to 144 Hours Postdose (AUC [0-144]) | Up to 144 hours postdose
  AUC (0-144) is defined as AUC from time 0 to 144 hours postdose, calculated by linear-linear trapezoidal summation.
Area Under the Analyte Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration (AUC [0-last]) | Up to Day 29
  AUC (0-last) is defined as AUC from time 0 to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Analyte Concentration-time Curve From Time Zero to Infinity (AUC [0-infinity]) | Up to Day 29
  AUC (0-infinity) is defined as AUC from time 0 to infinity, calculated as the sum of AUC (0-last) and C(last)/lambda(z); where C(last) is the last observed measurable (non-BQL) concentration; and lambda(z) is apparent terminal elimination rate constant.
Total Apparent Oral Clearance (CL/F) | Up to Day 29
  CL/F is defined as total apparent oral clearance, calculated as dose/AUC (0-infinity).
Apparent Volume of Distribution (Vd/F) | Up to Day 29
  Vd/F is defined as apparent volume of distribution, calculated as dose/[lambda (z)*AUC (0-infinity)].
Apparent Terminal Elimination Rate Constant (Lambda[z]) | Up to Day 29
  Lambda(z) is defined as apparent terminal elimination rate constant, estimated by linear regression using the terminal log-linear phase of the log-transformed concentration vs time curve.
Apparent Terminal Elimination Half-life (t1/2) | Up to Day 29
  t1/2 is defined as apparent terminal elimination half-life, calculated as 0.693/lambda(z).
Percentage of JNJ-56136379 Excreted in Urine (Ae,%Dose) | Up to Day 7
  Ae,%Dose is defined as cumulative urinary recovery represented as a percentage of dose, calculated as 100*(Aetotal/Dose).
Renal Clearance (CLr) | Up to 144 hours postdose
  CLr is defined as renal clearance, calculated as Ae(0-144h)/AUC(144h).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 8 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - The Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency